CLINICAL TRIAL: NCT03878875
Title: Does Sound Conditioning Protect Against Temporary Hearing Damage
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19CX4979
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hearing Loss, Noise-Induced
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Noise Exposure: One group (16, 8f:8m) with previous exposure i.e. nightclubs ++
  Interventions: Diagnostic Test: Session One Test Battery; Diagnostic Test: Session Two Test Battery; Diagnostic Test: Session Three Test Battery
- Low Noise Exposure: Group (16, 8f:8m) with less exposure measured through NESI
  Interventions: Diagnostic Test: Session One Test Battery; Diagnostic Test: Session Two Test Battery; Diagnostic Test: Session Three Test Battery

INTERVENTIONS:
Diagnostic Test: Session One Test Battery — Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (Around 35 minutes with breaks if required)
  * Extended Frequency Audiometry (~ 8 min), 0.25-16 kHz: Participants will be asked to press the button when they hear a sound through the headphones in a soundproof booth.
  * DPOAE (~ 5 min), 0.5-10 kHz: A small tip will be placed in participants' ear and they will hear a sound. The tip measures a response from hair cells in the cochlea and they will not need to do anything.
  * MEMR (~ 8 min), 4 kHz: A small tip placed in both ears and again a sound heard, however, this sound will gradually get louder until an involuntary muscle reflex is noted.
  * Speech-in-Noise Test (~ 5 min): Participants asked to repeat back a list of words as best as they can.
  * Tinnitus: Participants were also asked if they experience any tinnitus i.e. bilateral, lasting > 5 minutes. This was reported as Y/N.
Diagnostic Test: Session Two Test Battery — Exposure at single loud music event (Important that this is part of participants' normal recreational routine, and specifically require that attendance is not prompted by participation in this study): Participants to use sound level meter provided from the Audiology Department at Charing Cross Hospital or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session one - Ideally as soon as event is over.
Diagnostic Test: Session Three Test Battery — 1 week later (recovery): Repeat test battery.

SUMMARY:
This research project will contribute to the research surrounding the effect on the ear after noise exposure. This ever-growing field of research has never been more applicable than now with the increase of recreational noise exposure. Noise is the leading cause of preventable hearing loss and excessive occupational noise along with recreational noise exposure can cause a devastating disability. The World Health Organisation (WHO) estimates 1.1 billion young people could be at risk of hearing loss due to unsafe listening practices.

One of the mechanisms that could increase the resistance against noise induced hearing loss is 'sound conditioning'. Animal studies have found that prior exposure to low level noise over a period of a few weeks can 'condition' the ear. This conditioning then reduces the susceptibility to high level exposure i.e. strengthening the ear. In this study, the investigators aim to determine whether previous exposure to loud noise can condition the human ear, reducing the temporary hearing loss and temporary tinnitus ("ringing in the ear") that sometimes occurs after attending a loud nightclub or live music event.

There are many implications of this research. The long-term effects of non-damaging lifetime noise exposures are unclear. Principally, this research will allow better understanding about noise susceptibility and resistance, allowing for appropriate interventions, thus improving care. For instance, an individual more susceptible due to low prior exposure can be advised of risks and encouraged to use hearing protection. This thesis will increase the knowledge base surrounding the impacts of noise on hearing and educate others in understanding these.

DETAILED DESCRIPTION:
Objective: This study explored if sound conditioning (recent noise exposure) protects individuals against temporary hearing damage.

Design: Participants attended two sessions in this between-group repeated measures trial; the first included a noise exposure structured interview. Five dependent variables were measured before and after attending a loud event: EFA, DPOAE, MEMR, QuickSIN and Tinnitus. It was hypothesised those with high recent noise exposure, Group 1 (noise unit > 0.323), would experience less temporary hearing damage than irregular attendees, Group 0.

Sample: Thirty-two normal hearing participants with a mean age of 26 ± 3.3 years (16 males, 16 females).

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old (as age can affect cochlea hair cell function)
* Healthy participants with no significant medical conditions
* 0.25 Hz to 8 kHz PTA <= 20 dB HL indicating normal hearing
* Otoscopy to ensure no otological abnormalities
* No exposure to abnormally loud sounds in the past 24 hours
* Full capacity to consent
* Able to speak fluent English so information sheets, consent forms and instructions are fully understood
* Previous intention to attend a loud noise event during the course of the study, without the use of hearing protection

Exclusion Criteria:

* No permanent tinnitus or hyperacusis (sensitivity to loud sounds) which would mean participants are unable to undertake all testing and a high exposure event
* Any contraindications for testing i.e. excessive wax, infections
* One or more frequencies 0.25 Hz to 8 kHz > 20 dB HL in either ear
* Not involved in current research or have recently been involved in any research prior to recruitment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 32 Normal Hearing, Healthy 18-35-year-olds.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Frost, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Noise Exposure: One group with previous exposure i.e. nightclubs ++
  Session One Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test, Tinnitus Functional Index (Around 35 minutes with breaks if required)
  Session Two Test Battery: Exposure at single loud music event (Important that this is part of participants' normal recreational routine, and specifically require that attendance is not prompted by participation in this study): Participants to use sound level meter provided from the Audiology Department at Charing Cross Hospital to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session one - Ideally as soon as event is over.
  Session Three Test Battery: 1 week later (recovery): Repeat test battery.
- Low Noise Exposure: Group with less exposure measured through NESI
  Session One Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test, Tinnitus Functional Index (Around 35 minutes with breaks if required)
  Session Two Test Battery: Exposure at single loud music event (Important that this is part of participants' normal recreational routine, and specifically require that attendance is not prompted by participation in this study): Participants to use sound level meter provided from the Audiology Department at Charing Cross Hospital to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session one - Ideally as soon as event is over.
  Session Three Test Battery: 1 week later (recovery): Repeat test battery.
Period: Overall Study
Arm/Group | High Noise Exposure | Low Noise Exposure
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 participants in each group (0 and 1) tested across sessions.
Groups:
- High Noise Exposure; Low Noise Exposure: Session 1 Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (~35min with breaks if req)
  EFA (~8min), 0.25-16 kHz: Participants will be asked to press the button when they hear a sound through the headphones in a soundproof booth.
  DPOAE (~5min), 0.5-10 kHz: Small tip will be placed in participants' ear and they will hear a sound. The tip measures a response from hair cells in the cochlea and they will not need to do anything.
  MEMR (~8min), 4 kHz: A small tip placed in both ears and again a sound heard, however, this sound will gradually get louder until an involuntary muscle reflex is noted.
  Speech-in-Noise Test (~5min): Participants asked to repeat back a list of words as best as they can.
  Tinnitus: Participants were also asked if they experience any tinnitus i.e. bilateral, lasting >5min. Reported as Y/N
  Session 2: Exposure at single loud music event (Important that this is part of participants' normal recreational routine, and specifically require that attendance is not prompted by participation in this study): Participants to use sound level meter provided from the Audiology Department at Charing Cross Hospital or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session 1 - Ideally as soon as event is over.
  Session 3: 1 week later (recovery): Repeat test battery.
- Total: Total of all reporting groups
Arm/Group | High Noise Exposure | Low Noise Exposure | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: PTA (EF)
Description: Extended Frequency (EF) PTA with results measured in dBHL where higher values mean worse hearing thresholds.
  Hearing thresholds were measured in the two sessions (unfortunately session three was not completed). A single dB HL value was calculated by averaging results across participants in each session (Extended frequency audiometry (EFA) comprised of averaging 2-16 kHz).
Time Frame: 35 minutes per session
Population: For all parametric measures, participants were grouped into exposure and regression analysis assessed the group effect on the dependent variable. A range of categorical and continuous independent variables were controlled for against the dependent variable. Session three was excluded and not collected due to COVID-19.
Measure: Mean (Standard Deviation); unit: dB HL
Groups:
- High Noise Exposure; Low Noise Exposure: Session 1 Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (~35min with breaks if req)
  EFA (~8min), 0.25-16 kHz: Participants will be asked to press the button when they hear a sound through the headphones in a soundproof booth.
  Session 2: Exposure at single loud music event where participants used a sound level meter or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session 1 - Ideally as soon as event is over.
Arm/Group | High Noise Exposure | Low Noise Exposure
Number analyzed (Participants) | 16 | 16
dB HL
  Session 1 | 7.06 (8.15) | 8.94 (5.46)
  Session 2 | 7.94 (8.35) | 12.19 (6.45)
Statistical Analysis 1: Comparison: High Noise Exposure vs Low Noise Exposure; Test type: Superiority — Multiple linear regressions analysed the effect of conditioning (group) on each outcome at the second time point - session 2 (after noise exposure), controlling for session 1 outcome (before noise exposure), event exposure, age, and gender. It was hypothesised those with high recent noise exposure, Group 1 (noise unit > 0.323), would experience less temporary hearing damage than irregular attendees, Group 0; p < 0.0005, Regression, Linear; Group coefficient = -2.153; F(5, 26) = 116.044

2. Primary Outcome: DPOAE (DP)
Description: Distortion Product Otoacousic Emissions (DPOAE), DPOAEs were recorded bilaterally (at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 10 kHz) using the Otometrics Madsen Capella2. A daily check was performed in a 2 cc test cavity and tester's own ear to verify suitable recordings and ensure the probe was providing true responses. Measure results in the two sessions (unfortunately session three was not completed). DPOAE measurements were separated into distortion product (DP - dB SPL) and signal-to-noise ratio (SNR - dB) and averaged from 2-10 kHz. A single value was calculated by averaging results across participants in each session.
Time Frame: 35 minutes per session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB SPL
Groups:
- High Noise Exposure; Low Noise Exposure: Session 1 Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (~35min with breaks if req)
  DPOAE (~5min), 0.5-10 kHz: Small tip will be placed in participants' ear and they will hear a sound. The tip measures a response from hair cells in the cochlea and they will not need to do anything.
  Session 2: Exposure at single loud music event where participants used a sound level meter or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session 1 - Ideally as soon as event is over.
Arm/Group | High Noise Exposure | Low Noise Exposure
Number analyzed (Participants) | 16 | 16
dB SPL
  DP (2-10 kHz), Session 1 | 1.25 (5.03) | -0.06 (4.86)
  DP (2-10 kHz), Session 2 | 1.75 (5.04) | -0.88 (4.53)
Statistical Analysis 1: Comparison: High Noise Exposure vs Low Noise Exposure; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0005, Regression, Linear; Group coefficient = 1.602; F(5, 26) = 12.839

3. Primary Outcome: DPOAE (SNR)
Description: as for outcome 2
Time Frame: 35 minutes per session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | High Noise Exposure | Low Noise Exposure
Number analyzed (Participants) | 16 | 16
dB
  SNR (2-10 kHz), Session 1 | 12.94 (4.33) | 11.63 (4.15)
  SNR (2-10 kHz), Session 2 | 13.13 (4.63) | 11.19 (3.85)
Statistical Analysis 1: Comparison: High Noise Exposure vs Low Noise Exposure; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0005, Regression, Linear; Group coefficient was 1.059; F(5, 26) = 8.391

4. Primary Outcome: MEMR
Description: Middle Ear Muscle Reflex (MEMR) measured at 4 kHz bilaterally in dB SPL. A reflex was defined as > 0.02 ml compliance with appropriate morphology free from artefacts. Measure if MEMR is present/raised in the sessions. Averages between ears were also calculated for MEMR to give one result per participant for each session. A single value was then calculated by averaging results across participants in each session.
Time Frame: 35 minutes per session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB SPL
Groups:
- High Noise Exposure; Low Noise Exposure: Session 1 Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (~35min with breaks if req)
  MEMR (~8min), 4 kHz: A small tip placed in both ears and again a sound heard, however, this sound will gradually get louder until an involuntary muscle reflex is noted.
  Session 2: Exposure at single loud music event where participants used a sound level meter or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session 1 - Ideally as soon as event is over.
Arm/Group | High Noise Exposure | Low Noise Exposure
Number analyzed (Participants) | 16 | 16
dB SPL
  Session 1 | 88.91 (7.41) | 88.44 (8.56)
  Session 2 | 91.25 (6.71) | 90.31 (10.20)
Statistical Analysis 1: Comparison: High Noise Exposure vs Low Noise Exposure; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Regression, Linear; Group coefficient was 0.635; F(5, 26) = 6.416

5. Primary Outcome: SiN
Description: Speech in Noise (SiN) Test, Score. The sound field JBL Control One speakers and the Kamplex KM4 sound level meter (SLM) were calibrated via Guymark. Daily checks were conducted to assess speaker reliability when administering QuickSIN (Etymotic Research, 2001) with the signal and noise presented from the same speaker at 0° azimuths. The SLM confirmed speaker calibration and sound levels presented were within tolerances. Measure SiN in the sessions and a single value was calculated by averaging results across participants in each session.
Time Frame: 35 minutes per session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Groups:
- High Noise Exposure; Low Noise Exposure: Session 1 Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (~35min with breaks if req)
  Speech-in-Noise Test (~5min): Participants asked to repeat back a list of words as best as they can.
  Session 2: Exposure at single loud music event where participants used a sound level meter or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session 1 - Ideally as soon as event is over.
Arm/Group | High Noise Exposure | Low Noise Exposure
Number analyzed (Participants) | 16 | 16
dB
  Session 1 | 2.38 (2.53) | 2.94 (2.77)
  Session 2 | 1.38 (2.73) | 2.44 (2.76)
Statistical Analysis 1: Comparison: High Noise Exposure vs Low Noise Exposure; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Regression, Linear; Group coefficient was -0.383; F(5, 26) = 5.805

6. Primary Outcome: Tinnitus
Description: Participants were also asked if they experience any tinnitus i.e. bilateral, lasting > 5 minutes. This was reported as Y/N. An increase in underlying tinnitus, no change in underlying tinnitus and newly reported tinnitus was counted for each group in the second session. We aimed to assess the effect of conditioning on tinnitus change (i.e. increasing or not) at session 2, adjusting for tinnitus reported at session 1, age, gender, and event exposure. Session 1: existing underlying tinnitus reported. Session 2: Newly reported tinnitus and increase in underlying tinnitus.
Time Frame: 35 minutes per session
Population: Session three was excluded and not collected due to COVID-19.
Measure: Number; unit: participants
Groups:
- High Noise Exposure; Low Noise Exposure: Session 1 Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (~35min with breaks if req)
  Tinnitus: Participants were also asked if they experience any tinnitus i.e. bilateral, lasting >5min. Reported as Y/N
  Session 2: Exposure at single loud music event where participants used a sound level meter or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session 1 - Ideally as soon as event is over.
Arm/Group | High Noise Exposure | Low Noise Exposure
Number analyzed (Participants) | 16 | 16
participants
  Session 1 | 5 | 1
  Session 2 | 5 | 7
Statistical Analysis 1: Comparison: High Noise Exposure vs Low Noise Exposure; Test type: Superiority — A binary logistic regression was employed to assess the effect of conditioning on tinnitus change (i.e. increasing or not) at session 2, adjusting for tinnitus reported at session 1, age, gender, and event exposure; p < 0.005, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.071 to 1.85], Standard Error of Mean 0.140

ADVERSE EVENTS:
Time Frame: 3 months
Description: Any questions concerning adverse event reporting should be directed to the Principal Investigator. An SAE form should be completed within 24 hours. However, and hospitalisations for elective treatment of a pre-existing condition do not need reporting as SAEs. 'related', ie resulted from the administration of any of the research procedures; and 'unexpected', ie an event that is not listed in the protocol as an expected occurrence. This study did not put participants at risk.
Groups:
- High Noise Exposure (16, 8f:8m); Low Noise Exposure (16, 8f:8m): Session One Test Battery: Prior to noise exposure:
  Test battery - High-frequency audiometry, Distortion Product Otoacoustic Emissions, Middle Ear Muscle Reflex, Speech-in-Noise test (Around 35 minutes with breaks if required)
  Extended Frequency Audiometry (~ 8 min), 0.25-16 kHz: Participants will be asked to press the button when they hear a sound through the headphones in a soundproof booth.
  DPOAE (~ 5 min), 0.5-10 kHz: A small tip will be placed in participants' ear and they will hear a sound. The tip measures a response from hair cells in the cochlea and they will not need to do anything.
  MEMR (~ 8 min), 4 kHz: A small tip placed in both ears and again a sound heard, however, this sound will gradually get louder until an involuntary muscle reflex is noted.
  Speech-in-Noise Test (~ 5 min): Participants asked to repeat back a list of words as best as they can.
  Session Two Test Battery: Exposure at single loud music event (Important that this is part of participants' normal recreational routine, and specifically require that attendance is not prompted by participation in this study): Participants to use sound level meter provided from the Audiology Department at Charing Cross Hospital or sound level meter applications to measure sound levels inside the loud event.
  Morning after exposure: Repeat test battery from session one - Ideally as soon as event is over.
  Session Three Test Battery: 1 week later (recovery): Repeat test battery.
Arm/Group | High Noise Exposure (16, 8f:8m) | Low Noise Exposure (16, 8f:8m)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Session 3 was excluded and incomplete due to retention, unavailability of testing rooms resulting from COVID-19 and participants attending loud events after session 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03878875/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03878875/ICF_000.pdf